CLINICAL TRIAL: NCT03768427
Title: A Phase 3 Randomized, Active-comparator-controlled Clinical Study to Evaluate the Efficacy and Safety of Ezetimibe/Atorvastatin Combination Tablet (MK-0653C) as Second Line Lipid Lowering Treatment in Chinese Participants
Brief Title: Ezetimibe (EZ)/Atorvastatin (Ator) (MK-0653C) vs. Ator in Chinese Hypercholesterolemic Participants (MK-0653C-439)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653C-439; MK-0653C-439 (Other: Merck Protocol Number)
Record Dates: First submitted 2018-11-29; First posted 2018-12-07 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2023-04

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- EZ 10 mg/Ator 10 mg (Experimental): Single oral dose of EZ10mg/Ator10mg FDC tablet once daily (QD) for 84 days
  Interventions: Combination Product: EZ 10 mg/Ator 10 mg; Drug: Placebo for FDC EZ/Ator
- Atorvastatin 20 mg (Active Comparator): 2 atorvastatin 10 mg tablets administered orally, QD for 84 days
  Interventions: Drug: Atorvastatin; Drug: Placebo for atorvastatin
- EZ 10 mg/Ator 20 mg (Experimental): Single oral dose of EZ10mg/Ator20mg FDC tablet QD for 84 days
  Interventions: Combination Product: EZ 10 mg/Ator 20 mg; Drug: Placebo for FDC EZ/Ator
- Atorvastatin 40 mg (Active Comparator): 2 atorvastatin 20 mg tablets administered orally, QD for 84 days
  Interventions: Drug: Atorvastatin; Drug: Placebo for atorvastatin

INTERVENTIONS:
Combination Product: EZ 10 mg/Ator 10 mg — FDC of EZ10 mg/Ator 10mg
  Arms: EZ 10 mg/Ator 10 mg
Combination Product: EZ 10 mg/Ator 20 mg — FDC of EZ10 mg/Ator 20mg
  Arms: EZ 10 mg/Ator 20 mg
Drug: Atorvastatin — Atorvastatin administered orally QD, either as two 10 mg tablets or as two 20 mg tablets
  Other Names: Lipitor^®
  Arms: Atorvastatin 20 mg; Atorvastatin 40 mg
Drug: Placebo for FDC EZ/Ator — A single placebo tablet administered orally QD for 84 days
  Arms: EZ 10 mg/Ator 10 mg; EZ 10 mg/Ator 20 mg
Drug: Placebo for atorvastatin — Two placebo tablets matching atorvastatin administered orally QD for 84 days
  Arms: Atorvastatin 20 mg; Atorvastatin 40 mg

SUMMARY:
This study will evaluate the EZ/Ator fixed-dose combination (FDC) tablet (MK-0653C) as second line Low-Density Lipoprotein - Cholesterol (LDL-C) treatment in Chinese participants. The primary hypothesis is that MK-0653C 10/10 mg is superior to atorvastatin 20 mg in percent change from baseline in LDL-C to 12 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Has hypercholesterolemia diagnosed by investigator according to Chinese Guidelines on Prevention and Treatment of Dyslipidemia in Adults (2016 Edition).
* Has been stabilized on atorvastatin treatment at 10 mg or 20 mg (or other statins with LDL-C lowering efficacy equivalent to atorvastatin) for at least 4 weeks prior to Visit 1.
* If female, is not pregnant or breastfeeding, and is either not a woman of childbearing potential (WOCBP), or is a WOCBP who has used a contraceptive consistent with local regulations.
* If male, has used a contraceptive consistent with local regulations.
* Agrees to maintain a stable diet and stable exercise during the study.

Exclusion Criteria:

* Has uncontrolled hypertriglyceridemia which needs drug intervention or a fasting triglyceride (TG) value ≥500 mg/dL (4.52 mmol/L).
* Is currently treated with statin at dose of equivalent LDL-C lowering effect >20 mg atorvastatin.
* Has active liver disease
* Has New York Heart Association (NYHA) Class III or IV symptomatic congestive heart failure at Visit 1.
* Has had uncontrolled cardiac arrhythmias, myocardial infarction, percutaneous coronary intervention, coronary artery bypass graft, unstable angina, or stroke within 3 months (12 weeks) prior to Visit 1.
* Has homozygous familial hypercholesterolemia or has undergone LDL apheresis.
* Has endocrine or metabolic disease known to influence serum lipids or lipoproteins (i.e., secondary causes of hyperlipidemia, e.g., hyper or hypothyroidism, Cushing's syndrome).
* Has had a gastrointestinal tract bypass, or other significant intestinal malabsorption.
* Has a history of cancer within the past 5 years from Visit 1 (except for successfully treated dermatological basal cell or squamous cell carcinoma or in situ cervical cancer).
* Is known to be human immunodeficiency virus (HIV) positive.
* Has hypersensitivity or intolerance to ezetimibe, atorvastatin, the ezetimibe/atorvastatin combination tablet, or any component of these medications or has a condition or situation, which is described as a contraindication in labeling of EZETROL or Lipitor or may interfere with participation in the study.
* Has disorders of the hematologic, digestive, or central nervous systems including cerebrovascular disease and degenerative disease that would limit study evaluation or participation.
* Has a history of mental instability, drug/alcohol abuse within the past 5 years, or major psychiatric illness not adequately controlled and stable on pharmacotherapy.
* Has a history of myopathy or rhabdomyolysis with ezetimibe or any statin.
* Is a WOCBP who has had a positive urine pregnancy test within 24 hours before the first dose of study intervention. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Is currently taking medications that are potent modulators of cytochrome P-450 3A4 (CYP3A4) including: cyclosporine, systemically administered azole antifungals (e.g., ketoconazole, fluconazole, and itraconazole), macrolide antibiotics (e.g., clarithromycin, and erythromycin), protease inhibitors (e.g., ritonavir, saquinavir, and lopinavir), grapefruit or juice of grapefruit (200 ml/day for >3 times per week)
* Is taking any cyclical hormones (e.g., cyclical oral contraceptives, cyclical hormone replacement), including the combination of ethinyl estradiol and norethisterone, or non-cyclical hormones, including non-cyclical hormone replacement therapy (HRT) or any estrogen antagonist/agonist within 8 weeks.
* Note: If participant has been treated with a stable regimen of non-cyclical HRT for > 8 weeks and agree to continue this regimen for the duration of the trial, concomitant therapy is acceptable.
* Is receiving treatment with systemic corticosteroids (intravenous, intramuscular and oral steroids).
* Is treated with psyllium, other fiber-based laxatives, phytosterol margarine, and herbal medicine and/or over the counter (OTC) therapies that are known to affect serum lipids.
* Note: If participant has been treated with a stable regimen for > 8 weeks and agrees to continue this regimen for the duration of the trial, concomitant therapy is acceptable.
* Is treated with an anti-obesity drug (e.g. mazindol) within 12 weeks prior to Visit 1.
* Is treated with warfarin or warfarin-like anticoagulants and has not been on a stable dose with a stable International Normalized Ratio (INR) for at least 6 weeks.

weeks.

* Has taken lipid-lowering agents (except probucol) including, Cholestin, bile acid sequestrants, ezetimibe, fibrates or niacin (>200 mg/day), proprotein convertases subtilisin/kexin type 9 (PCSK9) inhibitors within 6 weeks prior to Visit 1.
* Has taken probucol within 10 weeks prior to Visit 1.
* Has been treated with any other investigational drug within 30 days.
* Currently follows an excessive weight reduction diet.
* Currently engages in a vigorous exercise regimen (e.g., marathon training, body building training) or intends to start training during the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (30):
- China (30):
  - The First Affiliated Hospital of Baotou Medical College ( Site 0025), Baotou, Anhui
  - Beijing Anzhen Hospital. Capital Medical University ( Site 0001), Beijing, Anhui
  - Aero Space center hospital ( Site 0003), Beijing, Beijing Municipality
  - Beijing Friendship Hospital ( Site 0005), Beijing, Beijing Municipality
  - Chongqing General Hospital ( Site 0037), Chongqing, Chongqing Municipality
  - Lanzhou University Second Hospital ( Site 0041), Lanzhou, Gansu
  - Guangdong General Hospital ( Site 0006), Guangzhou, Guangdong
  - The First Affiliated Hospital.Sun Yat-sen University ( Site 0007), Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital of Sun Yat-sen University ( Site 0008), Guangzhou, Guangdong
  - Daqing Oilfield General Hospital ( Site 0010), Daqing, Heilongjiang
  - The first affiliated Hospital of Harbin Medical University ( Site 0009), Haerbin, Heilongjiang
  - The Third Xiangya Hospital of Central South University ( Site 0013), Changsha, Hunan
  - Hunan Provincial People's Hospital ( Site 0011), Changsha, Hunan
  - Zhongda Hospital Southeast University ( Site 0045), Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University ( Site 0020), Nanjing, Jiangsu
  - First Affiliated Hospital of Soochow University ( Site 0048), Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University ( Site 0017), Xuzhou, Jiangsu
  - Subei People's Hospital ( Site 0040), Yangzhou, Jiangsu
  - Second Affiliated Hospital of Nanchang University ( Site 0038), Nanchang, Jiangxi
  - Ji Lin Province People Hospital ( Site 0016), Changchun, Jilin
  - China-Japan Union Hospital of Jilin University ( Site 0015), Changchun, Jilin
  - Central People s Hospital of Siping ( Site 0046), Siping, Jilin
  - The People's Hospital of Liaoning Province-Cardiovascular ( Site 0022), Shenyang, Liaoning
  - Zhongshan Hospital Fudan University ( Site 0049), Shanghai, Shanghai Municipality
  - Shanghai Tongji Hospital ( Site 0031), Shanghai, Shanghai Municipality
  - Tianjin Union Medicine Centre ( Site 0032), Tianjin, Tianjin Municipality
  - People s Hospital of Lishui City ( Site 0036), Lishui, Zhejiang
  - Ningbo First Hospital ( Site 0042), Ningbo, Zhejiang
  - Taizhou Hospital of Zhejiang Province ( Site 0035), Taizhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University ( Site 0034), Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qian J, Zhang X, Chen J, Ding C, Yang P, Qing L, Liu Y, Chen SS, Ge J. LDL-C Goal Attainment with Fixed-Dose Ezetimibe and Atorvastatin Versus High-Dose Atorvastatin in Chinese Patients: Subgroup Analysis of a Randomized Trial. Adv Ther. 2026 Jan 19. doi: 10.1007/s12325-025-03429-8. Online ahead of print. PMID 41553712
- [Derived] Qian J, Li Z, Zhang X, Chen J, Ding C, Yang P, Liu Y, Shi M, Ren X, Ge J; Phase III Study Investigators. Efficacy and Tolerability of Ezetimibe/Atorvastatin Fixed-dose Combination Versus Atorvastatin Monotherapy in Hypercholesterolemia: A Phase III, Randomized, Active-controlled Study in Chinese Patients. Clin Ther. 2022 Oct;44(10):1282-1296. doi: 10.1016/j.clinthera.2022.08.013. Epub 2022 Sep 29. PMID 36182594

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Chinese participants with Hypercholesterolemia inadequately controlled with 10 mg or 20 mg atorvastatin (Ator) monotherapy were enrolled.
Groups:
- Atorvastatin 10 mg - Ezetimibe 10 mg/Ator 10 mg: Participants had a 5-week run-in of atorvastatin 10 mg once daily (QD). They then received a single oral dose of ezetimibe (EZ) 10 mg/Ator 10 mg fixed dose combination (FDC) tablet QD, and 1 placebo tablet matched to active atorvastatin tablet QD for 84 days.
- Atorvastatin 10mg - Atorvastatin 20 mg: Participants had a 5-week run-in of atorvastatin 10 mg QD. They then received 2 atorvastatin 20 mg tablets QD, and 1 placebo tablet matched to active atorvastatin tablet QD for 84 days.
- Atorvastatin 20 mg - EZ 10 mg/Ator 20 mg: Participants had a 5-week run-in of atorvastatin 20 mg QD. They then received a single oral dose of EZ 10 mg/Ator 20 mg FDC tablet QD, and 1 placebo tablet matched to active atorvastatin tablet QD for 84 days.
- Atorvastatin 20 mg - Atorvastatin 40 mg: Participants had a 5-week run-in of atorvastatin 20 mg QD. They then received 2 atorvastatin 20 mg tablets administered orally, QD, and 1 placebo tablet matched to active atorvastatin tablet QD for 84 days.
Period: Overall Study
Arm/Group | Atorvastatin 10 mg - Ezetimibe 10 mg/Ator 10 mg | Atorvastatin 10mg - Atorvastatin 20 mg | Atorvastatin 20 mg - EZ 10 mg/Ator 20 mg | Atorvastatin 20 mg - Atorvastatin 40 mg
Started | 88 | 89 | 137 | 140
Completed | 76 | 85 | 126 | 129
Not Completed | 12 | 4 | 11 | 11
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0
Not completed — Physician Decision | 3 | 2 | 4 | 4
Not completed — Withdrawal by Subject | 7 | 2 | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin 10 mg - Ezetimibe 10 mg/Ator 10 mg | Atorvastatin 10mg - Atorvastatin 20 mg | Atorvastatin 20 mg - EZ 10 mg/Ator 20 mg | Atorvastatin 20 mg - Atorvastatin 40 mg | Total
Number analyzed (Participants) | 88 | 89 | 137 | 140 | 454
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.4 (7.4) | 62.4 (8.5) | 59.4 (9.3) | 60.6 (10.3) | 60.9 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 38 | 34 | 46 | 161
  Male | 45 | 51 | 103 | 94 | 293
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 88 | 89 | 137 | 140 | 454
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 88 | 89 | 137 | 140 | 454
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Baseline Low-Density Lipoprotein Cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] | 95.5 (24.6) | 96.8 (25.9) | 96.2 (25.2) | 88.4 (21.9) | 91.9 (24.9)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in LDL-C at Week 12
Description: Participants had LDL-C levels assessed at baseline and after 12 weeks of study drug administration. The change from baseline was calculated.
Time Frame: Baseline (Day 1) and Week 12
Population: All randomized participants who took at least one dose of study treatment, and have at least one post treatment observation of the respective endpoint (Baseline and Week 12) during the treatment period.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Atorvastatin 10 mg - Ezetimibe 10 mg/Ator 10 mg | Atorvastatin 10mg - Atorvastatin 20 mg | Atorvastatin 20 mg - EZ 10 mg/Ator 20 mg | Atorvastatin 20 mg - Atorvastatin 40 mg
Number analyzed (Participants) | 67 | 77 | 114 | 116
Percent change | -24.7 (24.9) | -5.3 (22.5) | -23.3 (23.1) | -9.1 (18.2)
Statistical Analysis 1: Comparison: Atorvastatin 10 mg - Ezetimibe 10 mg/Ator 10 mg vs Atorvastatin 10mg - Atorvastatin 20 mg; This statistical analysis was performed by fitting a constrained longitudinal model adjusting for time and the interaction of time by treatment, and time by baseline disease risk category, including all participants with baseline data (88 participants in arm "Atorvastatin 10 mg - ezetimibe 10 mg/Ator 10 mg" and 89 participants in arm "Atorvastatin 10mg - Atorvastatin 20 mg"); Test type: Other — Difference in least squares mean; p < 0.001, Constrained longitudinal model; Mean Difference (Final Values) = -19.5, 95% CI 2-sided [-26.7 to -12.3]; Difference in least squares mean is Atorvastatin 10 mg - EZ 10 mg/Ator 10 mg minus Atorvastatin 10mg - Atorvastatin 20 mg
Statistical Analysis 2: Comparison: Atorvastatin 20 mg - EZ 10 mg/Ator 20 mg vs Atorvastatin 20 mg - Atorvastatin 40 mg; This statistical analysis was performed by fitting a constrained longitudinal model adjusting for time and the interaction of time by treatment, and time by baseline disease risk category, including all participants with baseline data (137 participants in arm "Atorvastatin 20 mg - EZ 10 mg/Ator 20 mg" and 140 participants in arm "Atorvastatin 20 mg - Atorvastatin 40 mg"); Test type: Other — Difference in least squares mean; p < 0.001, Constrained longitudinal model; Mean Difference (Final Values) = -15.9, 95% CI 2-sided [-21.0 to -10.7]; Atorvastatin 20 mg - EZ 10 mg/Ator 20 mg minus Atorvastatin 20 mg - Atorvastatin 40 mg

2. Secondary Outcome: Percentage of Participants With An Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Time Frame: Up to approximately 17 weeks
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Atorvastatin 10 mg - Ezetimibe 10 mg/Ator 10 mg | Atorvastatin 10mg - Atorvastatin 20 mg | Atorvastatin 20 mg - EZ 10 mg/Ator 20 mg | Atorvastatin 20 mg - Atorvastatin 40 mg
Number analyzed (Participants) | 88 | 89 | 137 | 140
Percentage of Participants | 31.8 | 34.8 | 55.5 | 47.9

3. Secondary Outcome: Number of Participants Who Discontinued From Study Treatment
Description: The number of participants who discontinued treatment over the 12-week treatment period was assessed.
Time Frame: Up to approximately 15 weeks
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Number of Participants
Arm/Group | Atorvastatin 10 mg - Ezetimibe 10 mg/Ator 10 mg | Atorvastatin 10mg - Atorvastatin 20 mg | Atorvastatin 20 mg - EZ 10 mg/Ator 20 mg | Atorvastatin 20 mg - Atorvastatin 40 mg
Number analyzed (Participants) | 88 | 89 | 137 | 140
Number of Participants | 9 | 5 | 13 | 15

ADVERSE EVENTS:
Time Frame: Up to 17 weeks
Description: Serious AEs and Other AEs are presented for all participants who received ≥1 dose of study medication. All-Cause Mortality is presented for all participants randomized.
Arm/Group | Atorvastatin 10 mg - Ezetimibe 10 mg/Ator 10 mg | Atorvastatin 10mg - Atorvastatin 20 mg | Atorvastatin 20 mg - EZ 10 mg/Ator 20 mg | Atorvastatin 20 mg - Atorvastatin 40 mg
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/89 | 1/137 | 0/140
Serious Adverse Events (participants affected / at risk) | 2/88 | 4/89 | 10/137 | 6/140
Other Adverse Events (participants affected / at risk) | 0/88 | 0/89 | 7/137 | 2/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin 10 mg - Ezetimibe 10 mg/Ator 10 mg (N=88) | Atorvastatin 10mg - Atorvastatin 20 mg (N=89) | Atorvastatin 20 mg - EZ 10 mg/Ator 20 mg (N=137) | Atorvastatin 20 mg - Atorvastatin 40 mg (N=140)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian granulosa cell tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin 10 mg - Ezetimibe 10 mg/Ator 10 mg (N=88) | Atorvastatin 10mg - Atorvastatin 20 mg (N=89) | Atorvastatin 20 mg - EZ 10 mg/Ator 20 mg (N=137) | Atorvastatin 20 mg - Atorvastatin 40 mg (N=140)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 7 (7) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/27/NCT03768427/Prot_SAP_000.pdf